CLINICAL TRIAL: NCT03726008
Title: The Effect of a Perinatal Health Promotion Program on the Different Levels of Gestational Hyperglycemic Women's Bio-psycho-social Features and Child Growth
Brief Title: The Effect of a Perinatal Health Promotion Program on the Different Levels of Gestational Hyperglycemic Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Since the project has been terminated and there is no funding to continue the clinical trial
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-SV(I)-20160055
Record Dates: First submitted 2017-12-26; First posted 2018-10-31 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2019-04

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive the perinatal health promotion program and regular prenatal care
  Interventions: Behavioral: Perinatal health promotion program and regular prenatal care
- Control group (No Intervention): The control group will receive the regular perinatal care

INTERVENTIONS:
Behavioral: Perinatal health promotion program and regular prenatal care — Regular prenatal care and perinatal health promotion program including health promotion during pregnant period, health promotion during the ritual of Tso-Yueh-Tzu, health promotion during postpartum period, newborn care
  Arms: Experimental group

SUMMARY:
Taiwan National Health Insurance system was launched in 1995 and the diagnosis and treatment for gestational diabetes mellitus were reimbursed. However, controversy regarding treatment and prevention programs for the other different levels of gestational hyperglycemia continues. Moreover, long-term follow-up studies for the impact of different levels of gestational hyperglycemia on women's perinatal consequences were not found. Thus, the purpose of the study, is to explore the effect of a perinatal health promotion program on three different levels of gestational hyperglycemic women's bio-psycho-social features and their offspring's development.

DETAILED DESCRIPTION:
The investigators will recruit 120 women with three different levels of gestational hyperglycemia and assign them to either experimental group (a total of 60 women of gestational hyperglycemia) or control group (a total of 60 women of gestational hyperglycemia). Data will be collected at the women's six-month gestation, hospitalization for childbirth, and six weeks, six months, and one year postpartum. The three-year study findings can demonstrate the consequences and risk factors for women with three different levels of gestational hyperglycemia to suffer from type 2 diabetes mellitus. In addition, the results can be taken as an evidence-based intervention for the perinatal health promotion program in preventing the gestational hyperglycemic women to suffer from type 2 diabetes mellitus and in decreasing the impact of gestational hyperglycemia on the development of the gestational hyperglycemic women's offspring.

ELIGIBILITY:
Inclusion Criteria:The woman who

* Is 20 years old or above.
* Has a positive test for gestational diabetes mellifluous with the 75% oral glucose tolerance test during 24~28 gestation.
* Has junior high or above educational level.
* Can speak Mandarin Chinese.
* Is Taiwanese residence.
* Plans to give a childbirth at the medical center.

Exclusion Criteria:The woman who

-Is immigrant.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant wemon
Enrollment: 120 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Changes of biological indicator | women's six-month gestational age, about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  Fasting blood glucose test

SECONDARY OUTCOMES:
Changes of maternal body weight | women's six-month gestational age, about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  Maternal body weight(weight in kilograms)
Changes of maternal height | women's six-month gestational age, about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  Maternal height(height in meters)
Changes of newborn body weight | about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  Newborn body weight (weight in grams)
Changes of newborn body length | about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  Newborn body length (length in centimeter)
Changes of newborn head circumference | about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  Newborn head circumference (length in centimeter)
Changes of newborn Apgar score | about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  The newborn Apgar score in 1 and 5 minutes.The test is generally done at 1 and 5 minutes after birth and may be repeated later if the score is and remains low. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
Health information of newborn | about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  The newborn's health status and complications.
Changes of diabetes management self-efficacy Scale | women's six-month gestational age, about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  The Diabetes Management Self-efficacy Scale(DMSES) measures the individual's efficacy expectations for engaging in 20 type 2 diabetes self-management activities (Bijl et al., 1999).
  The scale is scored according to a 1-5 point numerical scale indicating the level of efficacy expectation the respondent has for each item with higher scores indicating greater levels of self-efficacy.
Changes of postpartum stress | about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  The 62-item Hung Postpartum Stress Scale (Hung PSS) is a valid and reliable tool for assessing women's postpartum stress during the 42-day postpartum period.
  Exploratory factor analysis indicated three components of postpartum stress: concerns about maternal role attainment, body changes and lack of social support (Hung, 2007) The Cronbach's alpha of the Hung PSS was 0.95. On a five-point Likert scale rating from 1 (not at all) - 5 (always), women rated each item on how often stress was perceived during the postpartum period. The score for postpartum stress was derived by summing all ratings, resulting in potential scores between 62-310. Higher values indicated a higher level of stress.
Changes of depression | women's six-month gestational age, about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  The 18-item Taiwanese Depression Questionnaire(TDQ) is widely used to screen for depression in Taiwan. The TDQ is a culture-specific, self-administered questionnaire; its sensitivity and specificity have been measured as 0.89 and 0.92, respectively (Lee, Yang, Lai, Chiu, & Chau, 2000). Using a 4-point Likert scale (i.e., 0-3), participants indicated whether and how often they experienced each item. Total scores ranged from 0 to 54; higher scores indicated more severe depression symptoms. The values of Cronbach's α at the five time points were .82 to .90.
Changes of health status | women's six-month gestational age, about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  We used the 12 items Chinese Health Questionnaire(CHQ) to measure perinatal women's health status (developed by Cheng (1985) and verified by Chong and Wilkinson (1989). Responses used a 4-point Likert scale (1 = not at all; 4 = most of the time). Responses of 1 or 2 were recoded as "0," responses of 3 or 4 were recoded as "1," and a total score ranging from 0 to 12 was calculated by summing the ratings (Chong & Wilkinson, 1989). The CHQ's sensitivity and specificity have been measured as 91.9% and 66.7%, respectively (Chong & Wilkinson, 1989); in this study, values of Cronbach's α ranged from .64 to .75 at the five time points.
Changes of blood pressure | women's six-month gestational age, about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  Blood pressure(with systolic, and diastolic)
Changes of body mass index | women's six-month gestational age, about 2 days after hospitalization for childbirth, and six weeks after childbirth, six months after childbirth, and one year after childbirth.
  Body mass index (kg/m^2)
Basic information of maternal | women's six-month gestational age
  Women's age, education, occupation, family income, marriage, pregnancy and production history

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Chi Yu, Master, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin Dist, Taiwan